CLINICAL TRIAL: NCT04793711
Title: EpiCeram for Skin Protection in Healthcare Workers Using Personal Protective Equipment
Brief Title: EpiCeram for Skin Protection in Healthcare Workers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find willing participants.
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPE-01
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-06

CONDITIONS: Irritant Contact Dermatitis
Keywords: dermatitis; PPE; healthcare workers
MeSH Terms: conditions — Dermatitis, Irritant; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EpiCeram (Experimental): Open-Label, 3 (three) times per day, topical, to hands and face, for 28 days.
  Interventions: Device: EpiCeram

INTERVENTIONS:
Device: EpiCeram — protective emollient

SUMMARY:
This is an open-label study using a device currently prescribed by doctors. This means everyone involved in the study will know the name of the product, only one product will be used, and the U.S. Food and Drug Administration (FDA) has approved the sale of this product. Although this is called a device, the product is an emollient-type lotion.

Healthcare workers (HCW) often suffer from signs and symptoms of skin irritation, including pain, redness, roughness, dryness, cracking and itching due to the extensive use of personal protective equipment (PPE) such as masks and gloves. These are thought to be due to changes in the normal skin barrier function induced by repeated minor abrasion in the warm, moist environment induced by extensive use of PPE required at work. EpiCeram Controlled Skin Barrier Emulsion (EpiCeram) is a prescription skin barrier repair product containing ingredients designed to improve skin barrier function. However, EpiCeram has not previously been studied in people with skin irritation due to extensive use of PPE.

This study was terminated after 1 (one) subject was enrolled due to the inability to find willing participants.

DETAILED DESCRIPTION:
At the screening visit, the study will be explained, and the participant will have the opportunity to ask questions. If the participant decides to enroll, they will have to read, sign and date this Informed Consent Document. The study staff will take the participants pertinent medical history to evaluate eligibility. The participant will be asked about the kind of skin products they are using as well as about use of PPE. Visit 2 activities may be performed at the Screening visit.

Participants will return to the study site one (1) week later and 28-days later to have Photographs, Skin Function Testing, and Laboratory Testing performed. The participant will be asked to avoid applying any skin products (except make-up) to the skin for the following week and for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. HCW using PPE at least 6 hours/day, 4 days/week or, depending on shift work, 24 hours/week, for at least one (1) month
2. Men or women, any age
3. Overall skin irritation score of at least 4 on 0-10 scale where 0 = none and 10 = worst
4. Willing to stop use of any other emollient and lotion for one (1) week between screening and baseline visit and for the duration of the study.
5. Participant is willing to stop use of or not begin use of any topical corticosteroids, emollients and lotions to the hands and face for the duration of the trial.

Exclusion Criteria:

1. History of any skin disorder existing prior to March 1, 2020 characterized by chronic visible lesions or skin irritation symptoms including, but not limited to atopic dermatitis, eczema, moderate-severe acne, chronic dry skin and psoriasis.
2. Use of topical corticosteroids within one (1) month of baseline visit.
3. History of any significant medical condition that, in the opinion of the investigator, might put the subject at risk in this trial.
4. Participation in another clinical trial within 30 days or 5 half-lives of the study agent, whichever is longer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levy, MD, Study Director — Director of Clinical Development
Locations (1):
- Sun Valley Arthritis Center, Peoria, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EpiCeram: Open-Label, 3 (three) times per day, topical, to hands and face, for 28 days.
  EpiCeram: Barrier cream
Period: Overall Study
Arm/Group | EpiCeram
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Arm EpiCeram: Open-Label to all subjects, no randomization.
Arm/Group | Active Arm EpiCeram
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Overall Irritation Score [Mean (Standard Deviation); unit: units on a scale] | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Reported Outcome of Overall Skin Irritation Symptoms
Description: A subjective assessment by the subject of combined, overall irritation of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Active Arm Epiceram: Open-Label, single-arm no randomization
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | 1 [1 to 1]

2. Primary Outcome: Change in Patient Reported Outcome of Pain
Description: A subjective assessment by the subject of pain of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | -2 [-2 to -2]

3. Primary Outcome: Change in Patient Reported Outcome of Redness
Description: A subjective assessment by the subject of redness of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | 0 [0 to 0]

4. Primary Outcome: Change in Patient Reported Outcome of Dryness
Description: A subjective assessment by the subject of dryness of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | -1 [-1 to -1]

5. Primary Outcome: Change in Patient Reported Outcome of Cracking
Description: A subjective assessment by the subject of cracking of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | -1 [-1 to -1]

6. Primary Outcome: Change in Patient Reported Outcome of Roughness
Description: A subjective assessment by the subject of roughness of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | -1 [-1 to -1]

7. Primary Outcome: Change in Patient Reported Outcome of Itching
Description: A subjective assessment by the subject of itching of face and hands using an ordinal scale of 0-10 where 0 = none and 10 = worst
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
score on a scale | -1 [-1 to -1]

8. Secondary Outcome: Change in Surface Skin pH
Description: A portable pH meter together with a combination pH electrode was used to measure pH on skin. An increase in value indicates a better result.
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: unitless
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
unitless | 0.04 [0.04 to 0.04]

9. Secondary Outcome: Change in Transepidermal Water Loss on Skin
Description: A light source wand was used to measure the outcome on skin of the dominant hand. Values were measured from 0 to 80 grams of water per square meter per hour; where 0 is equal to a very low level of water loss and 80 is the highest amount of water loss measured. An decrease in value indicates improvement.
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: grams of water per square meter per hour
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
grams of water per square meter per hour | 14 [14 to 14]

10. Secondary Outcome: Change in Stratum Corneum Hydration on Skin
Description: A light source wand was used to measure the outcome on skin of the dominant hand. Values were measured from 0 to 80; where 0 is equal to a very low level of hydration and 80 is the highest amount of hydration measured. An increase in value indicates improvement.
Time Frame: Baseline to Day 28
Measure: Mean (Full Range); unit: arbitrary units
Arm/Group | Active Arm Epiceram
Number analyzed (Participants) | 1
arbitrary units | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Screening through Day 28
Groups:
- Active Arm EpiCeram: Open-Label, single-arm, no randomization
Arm/Group | Active Arm EpiCeram
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination of the study after one subject, limited results and analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04793711/Prot_SAP_001.pdf